CLINICAL TRIAL: NCT02789306
Title: Influence of Maintenance Therapy on Peri-implant Disease
Brief Title: Preventive Maintenance Therapy on Peri-implant Diseases
Acronym: PIMT
Status: Completed | Type: Observational
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Collaborators: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Alberto Monje, DDS, Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain
Other Study IDs: 18002909
Record Dates: First submitted 2016-05-23; First posted 2016-06-03 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Periimplantitis; Periodontal Disease
Keywords: Preventive therapy; Dental implants
MeSH Terms: conditions — Peri-Implantitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Peri-implantitis: Peri-implantitis' - Loss radiographic bone beyond the biological bone remodeling at baseline (after prosthesis delivery) from the implant neck
  * Early:> 4 mm probing depth; <25% radiographic bone loss
  * Moderate:> 6mm probing depth; <50% radiographic bone loss
  * Severa:> 8 mm probing depth; > 50% radiographic bone loss
  Interventions: Procedure: Epidemiological study on the incidence of peri-implantitis
- Healthy: No signs of inflammation and otherwise no bone loss beyond the biological bone remodeling
  Interventions: Procedure: Epidemiological study on the incidence of peri-implantitis

INTERVENTIONS:
Procedure: Epidemiological study on the incidence of peri-implantitis — Clinical and radiographic examination in the routine based protocol

SUMMARY:
In the field of periodontics, periodontal support therapy has proven to be essential in preventing the incidence or recurrence of periodontal diseases. The protocol is designed according to the risk profile of a patient. For example, in the presence of the history of periodontal therapy, subgingival microbiota containing large numbers of spirochetes and mobile rods can recolonize pockets 4-8 weeks after scaling. Similarly, routine maintenance of dental implants has been recommended to prudently avoid peri-implant inflammation, Indeed, the understanding of the nature of the tissue around the implant and its pattern of disease would be important to consider, even surpassing importance. Recently, a systematic review by our group has identified the importance of maintenance therapy around implants because it can help prevent about 3 times patient-level frequency peri-implantitis.

Henceforth, our primary goal was to study the influence in a cross-sectional study of the frequency of peri-implantitis patients according to their post-implant placement and corresponding prosthesis visits supportive peri-implant maintenance. As such, it will be shown:

1. What are the local and systemic factors affecting the appearance of peri-implantitis
2. The ideal frequency of supportive peri-implant maintenance in patients who do not develop peri-implant disease
3. What is the population of patients who come to supportive peri-implant maintenance after placement of dental implants

DETAILED DESCRIPTION:
Cross-sectional analysis that will include consecutive patients with dental implants (> 250) with at least 36 months depending upon placement of the prosthesis. a cross-sectional study calling patients to whom implants have placed them in two private practices (CICOM, Badajoz and Nart Clinica Dental, Barcelona, Spain) in the last 36 month to conduct clinical and radiographic study was performed. This procedure is justified because of the high frequency of peri-implant disease (30%) and since there is no predictable and effective treatment, only prevention can improve the success rate and functionality.

- Clinical examination

A previously examiner (AN) calibrated perform all clinical measurements. The following clinical parameters were measured at six sites per implant (mesiobuccal, buccal, distobuccal, distolingual, lingual and mesiolingual):

1. Presence of plaque is recorded as 0 (no) or 1 (presence)
2. Degree of gingival redness recorded as 0 (no) or 1 (presence)
3. Depth bag measured from the gingival margin to the base of the bag in mm;
4. clinical attachment level (CAL) by the number of exposed threads measured
5. Bleeding on probing (BOP) recorded as 0 (no) or 1 (presence)
6. Discharge is recorded as 0 (no) or 1 (presence)
7. keratinized gingiva (mm)

   * Radiographic parameters A previously calibrated examiner perform radiographic measurement from the neck of the implant in the mesial and distal aspect of the implants using a digitized periapical. The software used for measurements will be ImageJ (approved by the American National Institute for Research - 'NIH')

ELIGIBILITY:
Eligibility criteria:

* Inclusion criteria

  1. Patients between 18 and 80 years old
  2. Consecutive patients that received dental implants in the last 36 months
  3. Patients with partial edentulism
  4. No antibiotic in the last 2 months
  5. Non-smoking or smoking <10 cigarettes a day
* Exclusion Criteria

  1. Uncontrolled systemic diseases
  2. Implants because prosthetic characteristics can not be registered probing depth or attachment level appropriately
  3. Smoking> 10 cigarettes a day
  4. Pregnant patients
  5. Implants not placed in our center

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cross-sectional analysis that will include patients with dental implants (> 250) with at least 36 months depending upon placement of the prosthesis. This procedure is justified because of the high frequency of peri-implant disease (30%) and since there is no predictable and effective treatment, only prevention can improve the success rate and functionality.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2016-05; Primary Completion 2017-01-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of peri-implantitis | 12 months
  * 'Peri-implant health' - Absence of bleeding or inflammation
  * 'Peri-implant mucositis' - Presence of bleeding (inflammation) but without bone loss
  * 'Peri-implantitis' - Lost of radiographic bone from the implant neck
    * Early:> 4 mm probing depth; <25% radiographic bone loss
    * Moderate:> 6mm probing depth; <50% radiographic bone loss
    * Severe:> 8 mm probing depth; > 50% radiographic bone loss

SECONDARY OUTCOMES:
Compliance of patients | 12 months
  * Every three months - 'compliers'
  * Every 6 months - 'compliers'
  * Between 6-12 months - 'erratic'
  * Sporadically - 'erratic'
  * Never after placement of restoration - 'non compliers'
Local and systemic factors on peri-implantitis | 12 months
  1. Sex (M / H)
  2. Age (years)
  3. Presence of periodontal disease in remaining teeth (determined by attachment level, probing depth, radiographic bone loss and presence of bleeding and / or discharge). By severity it will be stratified into 3 groups according to the 2015 American Academy of Periodontology (AAP):
     * Mild: Probing depth 3-5mm; bone loss <15%
     * Moderate: Probing depth: 5-7mm; 15-30% bone loss
     * Severe: Probing depth:> 7 mm; bone loss> 30%
  By location it will be stratified into two groups:
  * Generalized:> 30%
  * Localized: <30%
    5. Diabetes (Yes / No - blood glucose level mg / dl) 6. History of periodontal disease (Yes / No) 7. Time from implant placement (always> 6months after restoration) 8. Location of the implant
  * Posterior maxilla (MP)
  * Anterior maxilla (MA)
  * Mandibular posterior (mp)
  * Mandibular anterior (ma)

CONTACTS AND LOCATIONS:
Locations (1):
- Florencio Monje Gil, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Monje A, Aranda L, Diaz KT, Alarcon MA, Bagramian RA, Wang HL, Catena A. Impact of Maintenance Therapy for the Prevention of Peri-implant Diseases: A Systematic Review and Meta-analysis. J Dent Res. 2016 Apr;95(4):372-9. doi: 10.1177/0022034515622432. Epub 2015 Dec 23. PMID 26701350
- [Derived] Monje A, Wang HL, Nart J. Association of Preventive Maintenance Therapy Compliance and Peri-Implant Diseases: A Cross-Sectional Study. J Periodontol. 2017 Oct;88(10):1030-1041. doi: 10.1902/jop.2017.170135. Epub 2017 May 26. PMID 28548886